CLINICAL TRIAL: NCT02449551
Title: Study of AZD6094 (Volitinib) in Advanced Gastric Adenocarcinoma Patients With MET Amplification as a Third-line Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-07-167
Record Dates: First submitted 2015-05-14; First posted 2015-05-20 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Advanced Gastric Adenocarcinoma
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Volitinib (Experimental): Volitinib 800 mg will be administered orally once a day for 21 days as one cycle.
  Interventions: Drug: Volitinib

INTERVENTIONS:
Drug: Volitinib — Volitinib is an orally available, potent, selective, small molecule c-MET inhibitor. Volitinib 800 mg will be administered orally once a day for 21 days as one cycle.
  Other Names: AZD6094

SUMMARY:
Volitinib is a potent and selective small molecule c-Met kinase inhibitor. Volitinib was found to inhibit c-Met kinase at the enzyme and cell levels with IC50s of 4 nM for both enzyme and Met phosphorylation in the cell. Consistent with its potent enzyme and cell activity, volitinib was found to inhibit cell growth in vitro against tumors with c-Met gene amplification in the absence of HGF stimulation with IC50s generally below 10 nM. It also potently inhibited HGF-stimulated cell proliferation against tumors with c-Met overexpression or carrying a HGF/c-Met autocrine loop.

This study is a single-arm, phase II study of votilinib in patients with advanced gastric adenocarcinoma harboring MET amplification as a third line treatment Volitinib 800 mg will be administered orally once a day for 21 days as one cycle.

To investigate the efficacy of volitinib in patients with advanced gastric adenocarcinoma harboring MET amplification.

DETAILED DESCRIPTION:
same as above

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Advanced gastric adenocarcinoma (including GEJ) that has progressed during or after second-line therapy.

   * Both fluoropyrimidine and platinum agent need to be contained in the prior chemotherapies
   * Prior adjuvant or neoadjuvant therapy is counted as 1 regimen, provided that disease progression occurs within 6 months after the completion of adjuvant or neoadjuvant therapy.
4. Have the presence of measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
5. Patients with MET amplification.
6. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
7. Eastern Cooperative Oncology Group performance status 0-1.
8. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
9. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

   * Haemoglobin ≥9.0 g/dL (transfusion allowed)
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * White blood cells (WBC) > 3 x 109/L
   * Platelet count ≥100 x 109/L (transfusion allowed)
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (does not include patients with Glibert's disease)
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
   * Serum creatinine ≤1.5 x institutional ULN
10. At least one measurable lesion that can be accurately assessed by imaging or physical examination at baseline and following up visits.
11. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1. for women of childbearing potential.
12. Provision of consent for mandatory biopsy at progression (fresh frozen will be mandatory if clinically feasible)
13. Provision of archival or fresh tissue sample at baseline (fresh frozen will be mandatory if clinically feasible)

Exclusion Criteria:

1. Are currently enrolled in, or discontinued within the last 21 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
2. Any previous treatment with MET inhibitors
3. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
4. HER2 positive patients (defined by HER2 3+ by immunohistochemistry or HER2 SISH +)
5. Patients unable to swallow orally administered medication.
6. Treatment with any investigational product during the last 21 days before the enrollment (or a longer period depending on the defined characteristics of the agents used).
7. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 3 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denusomab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
8. With the exception of alopecia, any ongoing toxicities (>Common Toxicity Criteria for Adverse Effects grade 1) caused by previous cancer therapy.
9. Intestinal obstruction or Common Toxicity Criteria for Adverse Effects grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
10. Resting ECG with measurable QTcB > 480 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
11. Patients with cardiac problem as follows: uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy) Baseline Left ventricular ejection fraction below the LLN of <55% measured by echocardiography or institution's LLN for MUGA, Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest , Symptomatic heart failure (NYHA grade II-IV), Prior or current cardiomyopathy, Severe valvular heart disease, Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy), Acute coronary syndrome within 6 months prior to starting treatment
12. Female patients who are breast-feeding or child-bearing and Male or female patients of reproductive potential who are not employing an effective method of contraception
13. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
14. Patients currently receiving (or unable to stop use at least 2 weeks) prior to receiving the first dose of AZD6094, medications known to be potent inhibitors of CYP1A2 or CYP3A4, potent inducers of CYP3A4 or CYP3A4 substrates with a narrow therapeutic range.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 8 weeks

SECONDARY OUTCOMES:
Objective response rate (ORR) | 8 weeks
Duration of response | 8 weeks
Disease control rate | 8 weeks
Overall survival (OS) | 8 weeks
Number of subjects with Adverse Events as a measure of safety and tolerability | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jee yun Lee, MD,Ph.D., Principal Investigator — Samsung Medical Center,Seoul,Korea
Locations (1):
- Samsung Medical center, Seoul, South Korea